CLINICAL TRIAL: NCT03737656
Title: Open-label, Randomized, Clinical Trial With Three Groups for the Characterization of Pharmacokinetics of a Vaginal Ring With 2.0 g Progesterone in Post-menopausal Women
Brief Title: Characterization of the Pharmacokinetics of a Vaginal Ring With 2.0 g Progesterone in Post-menopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Collaborators: Grünenthal, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRG-02-GRU/PK-PVR-01; 16-CI-19 039 043 (Registry Identifier: Comisión Federal para la Protección contra Riesgos Sanitarios (COFEPRIS) Mexico); HP8013-01 (Other: Grünenthal)
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Pharmacokinetics
Keywords: Progesterone; Vaginal ring

STUDY DESIGN:
Intervention Model Description: Single site, open-label, randomized, single-dose, with three groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progesterone Vaginal Ring (Group A) (Experimental): Insertion of the vaginal ring on Day 1 and continuous use until 91 days of treatment are completed. In this group, 28 participants will be included.
  Interventions: Drug: Progesterone vaginal ring
- Progesterone Vaginal Ring (Group B) (Experimental): Insertion of the vaginal ring on Day 1, removal for 2 hours on study Day 28, re-insertion on Day 28, and continuous use for 63 days until 91 days of treatment are completed. In this group, 6 participants will be included.
  Interventions: Drug: Progesterone vaginal ring
- Progesterone Vaginal Ring (Group C) (Experimental): Insertion of the vaginal ring on Day 1, removal for 4 hours on study Day 28, re-insertion on Day 28, and continuous use for 63 days until 91 days of treatment are completed. In this group, 6 participants will be included.
  Interventions: Drug: Progesterone vaginal ring

INTERVENTIONS:
Drug: Progesterone vaginal ring — Vaginal ring with 2.0 g progesterone (sustained-release over 90-days)
  Other Names: Progering (Trade Mark)

SUMMARY:
This is a single site, open-label, randomized, single-dose, Phase 1 study in post-menopausal women.

DETAILED DESCRIPTION:
The objective of the study is to characterize the pharmacokinetics of progesterone in post-menopausal women after the insertion of a vaginal ring containing 2.0 g of progesterone. Progesterone is slowly released from the ring within 90 days (sustained-release). Study participants will use the vaginal ring for a period of 91 days (13 weeks).

Progesterone blood concentrations will be determined during the use of the vaginal ring and after removal of the vaginal ring after a period of use of 13 weeks. In subgroups of participants, progesterone blood concentrations will also be determined after removal of the ring for a period of 2 hours or 4 hours on Day 28 of use. A study participant has completed the study when the final evaluation takes place, which is 7-15 days after removal of the vaginal ring on Day 91.

The safety of the progesterone vaginal ring will be assessed based on the adverse events reported.

ELIGIBILITY:
Inclusion Criteria:

A. Only post-menopausal women aged between 40 years and 65 years who are currently not in hormone replacement therapy and who meet any of the following criteria:

1. 12 months of spontaneous and continuous amenorrhea.
2. 6 months of spontaneous amenorrhea with follicle-stimulating hormone levels above 40 international units/liter and less than 20 picograms per milliliter estradiol.
3. Bilateral oophorectomy without hysterectomy.

B. The body mass index must be between 18.5 and 29.99 kilograms per square meter according to the Quetelet index.

C. Participants must be healthy determined by the results of a complete clinical history recorded by the clinical investigational site and the results of the laboratory examinations done by a certified clinical laboratory.

D. Participants with pre-existing illnesses must be controlled with stable doses of medication for a period of at least 3 months.

E. The allowed limits of variation within normal in the screening visit will be: systolic blood pressure (sitting) less or equal to 130 mmHg, diastolic blood pressure less or equal to 80 mmHg, pulse rate between 50 and 100 beats per minute for 1 minute and respiratory rate between 14 and 20 breaths per minute.

F. Laboratory and other examinations to be conducted for the inclusion of participants will be:

1. Complete blood count: leukocytes, erythrocytes, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, erythrocyte distribution width, platelets, neutrophils, lymphocytes, monocytes, eosinophils.
2. Blood chemistry 27 elements: glucose, urea, blood urea nitrogen (BUN), creatinine, BUN/creatinine ratio, uric acid, cholesterol, high-density lipoprotein (HDL) cholesterol, triglycerides, low-density lipoprotein cholesterol, non-HDL cholesterol, atherogenic index, total protein, albumin, globulins, albumin/globulin ratio, total bilirubin, direct bilirubin, indirect bilirubin, aspartate aminotransferase, alanine aminotransferase, total alkaline phosphatase, gamma-glutamyl transferase, lactate dehydrogenase, iron, calcium, sodium, potassium, and chloride.
3. Urinalysis: Physical examination (color, appearance, density); chemical examination (pH, leukocytes, nitrite, protein, glucose, ketones, bilirubin, urobilinogen, hemoglobin); microscopic examination (leukocytes, erythrocytes, dysmorphic erythrocytes, casts, crystals, squamous epithelial cells, tubular renal cells, mucus, bacteria and yeasts).
4. Hepatitis B screening (antibody to hepatitis B core antigen [Anti-HBc], antibody to hepatitis B surface antigen [HBs-Ab], antibody to hepatitis B surface antigen [Anti-HBs]) and hepatitis C antibodies.
5. HIV test: Antibodies to the human immunodeficiency virus (Anti-HIV 1 and 2).
6. Venereal disease research laboratory test (VDRL).
7. Drugs of abuse test at the screening visit and approximately 12 hours before insertion of the vaginal ring on Day 1.
8. Alcohol breath test approximately 12 hours before insertion of the vaginal ring on Day 1.
9. Twelve-lead electrocardiogram (ECG) (with validity of no more than 3 months). The ECG will be performed after resting for 5 minutes in a sitting position.
10. Gynecological profile:

    * Follicle-stimulating hormone.
    * Serum estradiol.
    * Luteinizing hormone.
11. Transvaginal ultrasound (without clinically significant findings).
12. Pap smear without clinically significant findings.
13. Bilateral mammography (with Breast Imaging Reporting and Data System [BI-RADS] 1 or 2 results).

Exclusion Criteria:

A. Participants who do not meet the inclusion criteria described in the above section.

B. Participants with a history of the following diseases: cardiovascular (myocardial infarction, not-controlled hypertension, thromboembolic, arterial or venous diseases), renal (kidney failure), hepatic (hepatitis, cholestatic jaundice, hepatic tumors, Dubin-Johnson syndrome, Rotor syndrome), muscular, metabolic, gastrointestinal including constipation, neurologic (cerebrovascular disease), endocrinological (not-controlled diabetes), hematopoietic or any type of anemia, history of toxic shock due to Staphylococcus, asthma, mental disorder (depression) or other organic abnormalities that are not appropriately controlled and that require a pharmacological treatment that could result in a drug interaction with the study medication. Women who have had muscular trauma within 21 days previous to the study will also be excluded.

C. Participants with uterine bleeding.

D. Participants with endometrial thickness equal to or greater than 7 millimeters as determined in the transvaginal ultrasound.

E. Participants with history of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer.

F. Hypersensitivity or allergy to the study medication.

G. Participants who have been exposed to medications known to be enzyme inducers or inhibitors or women who have taken potentially toxic medications within 72 hours previous to the start of each study period.

H. Participants undergoing hormone replacement therapy or taking thyroid hormones in the last 3 months.

I. Participants who have been hospitalized for any reason within 6 months prior to study start.

J. Participants who have taken investigational medicinal products from other investigations within 180 days (i.e., 6 months) prior to study start.

K. Participants who have smoked tobacco within 12 hours prior to study days 1, 28, and 91.

L. Participants who have donated or lost more than 450 milliliters of blood within 60 days prior to study start.

M. Participants with a history of drug abuse or alcoholism.

N. Participants requiring a special diet for any reason e.g., vegetarian.

O. Participants unable to understand the nature, objectives, and possible consequences of the study.

P. Evidence of the participant's uncooperativeness during the conduct of the study.

Q. Positive results for drugs of abuse (in urine) or alcohol breath tests.

R. Participants who are not registered in the Mexico Ministry of Health (Comisión Federal para la Protección contra Riesgos Sanitarios [COFEPRIS]) webpage.

S. Relationship of subordination between the participants and the investigators.

T. Sponsor or clinical site employees.

Discontinuation criteria:

Participants may be discontinued from the study at the discretion of the Clinic Director among others, because of the following reasons:

A. Safety and well-being of the participant.

B. Lack of adherence to the procedures and therefore non-compliance with the protocol.

C. Medical reasons: adverse reactions to the study medication classified as severe.

D. Recurring or intercurrent disease (not controlled).

E. Withdrawal of consent to participate in the study.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Progesterone pharmacokinetic parameters (AUC0-t) | Insertion of ring (Day 1) to removal of ring (Day 91) plus 24 hours
  In Groups A, B, and C, 3 blood samples will be obtained before the device is placed and 24 samples after placement of the device up to Day 91. Additional samples (6 samples in Group B and 8 samples in Group C) will be taken while the ring is removed/after the ring is re-inserted on Day 28. Eight blood samples will be taken from all participants (from Groups A, B, and C) within 24 hours after the ring is removed on Day 91. Plasma concentrations of progesterone will be determined using validated analytical methods. The baseline-corrected and uncorrected area under the plasma concentration-time curve from 0 to time t (AUC0-t) will be calculated.
Progesterone pharmacokinetic parameters (AUC0-inf) | Insertion of ring (Day 1) to removal of ring (Day 91) plus 24 hours
  In Groups A, B, and C, 3 blood samples will be obtained before the device is placed and 24 samples after placement of the device up to Day 91. Additional samples (6 samples in Group B and 8 samples in Group C) will be taken while the ring is removed/after the ring is re-inserted on Day 28. Eight blood samples will be taken from all participants (from Groups A, B, and C) within 24 hours after the ring is removed on Day 91. Plasma concentrations of progesterone will be determined using validated analytical methods. The baseline-corrected and uncorrected area under the plasma concentration-time curve from 0 to infinity (AUC0-inf) will be calculated.
Progesterone pharmacokinetic parameters (Cmax) | Insertion of ring (Day 1) to removal of ring (Day 91) plus 24 hours
  In Groups A, B, and C, 3 blood samples will be obtained before the device is placed and 24 samples after placement of the device up to Day 91. Additional samples (6 samples in Group B and 8 samples in Group C) will be taken while the ring is removed/after the ring is re-inserted on Day 28. Eight blood samples will be taken from all participants (from Groups A, B, and C) within 24 hours after the ring is removed on Day 91. Plasma concentrations of progesterone will be determined using validated analytical methods. The baseline-corrected and uncorrected maximum plasma concentration (Cmax) will be calculated.

SECONDARY OUTCOMES:
Progesterone pharmacokinetic parameters (Tmax) | Insertion of ring (Day 1) to removal of ring (Day 91) plus 24 hours
  In Groups A, B, and C, 3 blood samples will be obtained before the device is placed and 24 samples after placement of the device up to Day 91. Additional samples (6 samples in Group B and 8 samples in Group C) will be taken while the ring is removed/after the ring is re-inserted on Day 28. Eight blood samples will be taken from all participants (from Groups A, B, and C) within 24 hours after the ring is removed on Day 91. Plasma concentrations of progesterone will be determined using validated analytical methods. The time to achieve maximum plasma concentration (tmax) will be calculated.
Progesterone pharmacokinetic parameters (AUC%extr) | Insertion of ring (Day 1) to removal of ring (Day 91) plus 24 hours
  In Groups A, B, and C, 3 blood samples will be obtained before the device is placed; 24 samples after placement of the device up to Day 91. Additional samples (6 samples in Group B and 8 samples in Group C) will be taken while the ring is removed/after the ring is re-inserted on Day 28. Eight blood samples will be taken from all participants (from Groups A, B, and C) within 24 hours after the ring is removed on Day 91. Plasma concentrations of progesterone will be determined using validated analytical methods. The extrapolated area under the plasma concentration-time curve (AUC%extr) will be calculated based on AUC0-t and AUC0-inf.
Progesterone pharmacokinetic parameters (t1/2) | Insertion of ring (Day 1) to removal of ring (Day 91) plus 24 hours
  In Groups A, B, and C, 3 blood samples will be obtained before the device is placed and 24 samples after placement of the device up to Day 91. Additional samples (6 samples in Group B and 8 samples in Group C) will be taken while the ring is removed/after the ring is re-inserted on Day 28. Eight blood samples will be taken from all participants (from Groups A, B, and C) within 24 hours after the ring is removed on Day 91. Plasma concentrations of progesterone will be determined using validated analytical methods. The elimination half-time (t1/2) will be calculated.
Progesterone pharmacokinetic parameters (MRT) | Insertion of ring (Day 1) to removal of ring (Day 91) plus 24 hours
  In Groups A, B, and C, 3 blood samples will be obtained before the device is placed; 24 samples after placement of the device up to Day 91. Additional samples (6 samples in Group B and 8 samples in Group C) will be taken while the ring is removed/after the ring is re-inserted on Day 28. Eight blood samples will be taken from all participants (from Groups A, B, and C) within 24 hours after the ring is removed on Day 91. Plasma concentrations of progesterone will be determined using validated analytical methods. The mean residence time (MRT) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (1):
- Investigacíon Farmacológica y Biofarmacéutica (IFaB), S.A.P.I. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Information available on the Grünenthal Web Site (see URL below for details)
Supporting Information: Study Protocol, SAP, CSR
URL: http://www.grunenthal.com/r-d-vision-mission/clinical-trials/data-sharing-clinical-trials